CLINICAL TRIAL: NCT02552017
Title: Accuracy of Detection Using ENdocuff Optimisation of Mucosal Abnormalities
Acronym: ADENOMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Tyneside and Sunderland NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 039/2014; 17718 (Registry Identifier: UK Clinical Research Network); 1182104 (Registry Identifier: International Standard Randomised Controlled Trial Number)
Record Dates: First submitted 2015-09-10; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Neoplasms; Colonic Polyps; Adenoma
Keywords: adenoma detection rate; Endocuff; Endocuff Vision; colonoscopy; bowel cancer screening; bowel cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps; Adenoma; Intestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endocuff Vision-assisted Colonoscopy (Active Comparator): Participants in this arm undergo Endocuff Vision-assisted colonoscopy
  Interventions: Device: Endocuff Vision
- Standard Colonoscopy (No Intervention): Participants in this arm undergo standard colonoscopy

INTERVENTIONS:
Device: Endocuff Vision — Endocuff Vision is a new device made of soft plastic material with a unique dynamic shape. It is manufactured by ARC Medical Design Limited and Diagmed in the United Kingdom. It has European Conformity in United Kingdom. The core is made of polypropylene and the 'finger like' projections are made of a thermoplastic elastomer. It comes in four colour coded sizes (purple, blue, green and orange) to fit a range of paediatric and adult colonoscopes. Endocuff Vision is the more updated version of device that has only one proximal row of more rounded finger-like projections. It is mounted at the tip of the colonoscope and held on by friction (pull-off force is a minimum of 10 Newtons).
  Arms: Endocuff Vision-assisted Colonoscopy

SUMMARY:
The purpose of this study is to determine if a new device, called the Endocuff Vision (a small plastic device attached to the end of the colonoscope which helps by holding the folds of the bowel back to give a clear view of the inside of the bowel) will significantly improve the detection of adenomas when used in all patients referred for colonoscopy.

DETAILED DESCRIPTION:
Bowel cancer is common in the United Kingdom, with around 1 in 16 men and 1 in 20 women developing it at some point in their lives. Most bowel cancers happen when a type of polyp (a growth in the bowel) called an adenoma becomes cancerous. Doctors use a camera test, known as a colonoscopy, to look inside the bowel and find these polyps and remove them. Removing precancerous polyps is known to reduce the chances of a person developing bowel cancer in the future. How good colonoscopists are at finding these polyps varies, and there is a lot of research into how to improve "adenoma detection rates".

A new device, called the Endocuff Vision (a small plastic device attached to the end of the colonoscope which helps by holding the folds of the bowel back to give a clear view of the inside of the bowel) has been shown to improve the rate of polyp detection at colonoscopy, and to make polyp removal easier. Previous small studies have shown that there is a significant improvement in detection of adenomas when an Endocuff Vision is used (with the rate of detection of adenomas rising from 49% to 66%). Colonoscopists who have used the Endocuff Vision before also feel that polyp removal is easier when it is on the colonoscope. This study will randomise patients coming for colonoscopy to have their procedure performed as usual (i.e. without the Endocuff Vision attached) or as an Endocuff Vision-assisted colonoscopy. The investigators will record polyp and adenoma detection rates, duration of procedure, participant comfort levels, and complications. All patients referred for colonoscopy (via the symptomatic service, surveillance procedures, and the Bowel Cancer Screening Programme) will be invited in 7 centres (a mixture of specialist centres and district general hospitals), recruiting a total of 1772 participants.

ELIGIBILITY:
Inclusion Criteria:

1. All patients referred for screening, surveillance, or diagnostic colonoscopy
2. All patients must be able to give informed consent

Exclusion Criteria:

1. Patients with any absolute contraindications to colonoscopy
2. Patients with established or suspicion of large bowel obstruction or pseudo-obstruction
3. Patients with known colon cancer or polyposis syndromes
4. Patients with known colonic strictures
5. Patients with known severe diverticular segments (that is likely to impede colonoscope passage)
6. Patients with active colitis (ulcerative colitis, Crohn's colitis, diverticulitis, infective colitis)
7. Patients lacking capacity to give informed consent
8. Pregnancy
9. Patients who are on clopidogrel, warfarin, or other new generation anticoagulants who have not stopped this for the procedure.
10. Patients who are attending for a therapeutic procedure or assessment of a known lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1772 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 10 months
  A difference in adenoma detection rate between Endocuff Vision-assisted colonoscopy and standard colonoscopy.

SECONDARY OUTCOMES:
Mean adenomas detected per procedure | 10 months
  A difference in mean adenomas detected per procedure between both groups
Rate of cuff exchange | 10 months
  The rate of cuff exchange (that is, how often the cuff has to be removed) between both groups
Effect on duration of caecal intubation rates | 10 months
  Duration of complete withdrawal time in procedures where no polyps are detected between both groups
Patient satisfaction using validated patient comfort Bowel Cancer Screening Programme (BCSP) questionnaires | 10 months
  Patient satisfaction measured from no pain (0) to severe pain (3), episodes of discomfort from no discomfort (0) to frequent (more than 4 times)(3), length of discomfort from no discomfort (0) to more than 1 minute(3).
Increase in surveillance colonoscopies caused by increased adenoma detection rate | 10 months
  Increase in surveillance colonoscopies due to increased adenoma detection rate in terms of number of potential follow up procedures based on British Society of Gastroenterology adenoma surveillance guidelines in both groups
Number of proximal sessile serrated polyps by histology | 10 months
  Number of of proximal sessile serrated polyps in both groups
Polyp location | 10 months
  Distribution of polyps in the colon in both groups by location
Adenoma detection rate of BCSP and non-BCSP endoscopists | 10 months
  Adenoma detection rate of BCSP and non-BCSP colonoscopists
Change in adenoma detection rate of each endoscopist during the course of the trial | 10 months
  Adenoma detection rate (ADR) of the first 20% of patients scoped by each colonoscopist with the last 20% of patients in each arm to identify any changes in ADR.
Adenoma detection rate of individual endoscopist before and after trial commencement | 10 months
  Baseline ADR of each colonoscopist prior to trial recruitment with their individual ADR in patients where Endocuff Vision was not used.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Rees, MBBS, FRCP, Principal Investigator — South Tyneside and Sunderland NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - County Durham and Darlington NHS Foundation Trust, Durham, County Durham
  - North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees, County Durham
  - St Mark's Hospital and Academic Institute, Harrow, Middlesex
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough, North Yorkshire
  - Northumbria Healthcare NHS Foundation Trust, North Shields, Tyne and Wear
  - South Tyneside NHS Foundation Trust, South Shields, Tyne and Wear
  - City Hospitals Sunderland NHS Foundation Trust, Sunderland, Tyne and Wear

REFERENCES:
- [Derived] Ngu WS, Bevan R, Tsiamoulos ZP, Bassett P, Hoare Z, Rutter MD, Clifford G, Totton N, Lee TJ, Ramadas A, Silcock JG, Painter J, Neilson LJ, Saunders BP, Rees CJ. Improved adenoma detection with Endocuff Vision: the ADENOMA randomised controlled trial. Gut. 2019 Feb;68(2):280-288. doi: 10.1136/gutjnl-2017-314889. Epub 2018 Jan 23. PMID 29363535